CLINICAL TRIAL: NCT05799300
Title: A Retrospective, Observational, Single-centre, Cohort Database Analysis of the Haemodynamic Effects of Low-dose Spinal Anaesthesia for Hip Fracture Surgery.
Brief Title: Haemodynamic Effects of Low-dose Spinal Anaesthesia for Hip Fracture Surgery.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Sussex County Hospital (Other)
Responsible Party: Principal Investigator, Stuart White, Consultant Anaesthetist, Chief Investigator, Royal Sussex County Hospital
Other Study IDs: RoyalSussex
Record Dates: First submitted 2023-02-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Hip Fractures
Keywords: Anaesthesia, spinal; Anaesthesia, cardiovascular effects; Surgery, hip fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip fracture cohort: Gender, Age, Racial and Ethnic Origin of Subjects Male and female adults over the age of 18 years; all origins, all races will be included.
  Inclusion/exclusion criteria as below
  Interventions: Procedure: Intrathecal anaesthesia

INTERVENTIONS:
Procedure: Intrathecal anaesthesia — Low dose 0.5% hyperbaric bupivacaine (1.3mls, 0.65mg) intrathecal anaesthesia.

SUMMARY:
Approximately 65, 000 hip fractures occur in the United Kingdom (UK) each year, and more than 99% are repaired by surgery. Roughly half of patients receive spinal anaesthesia, where a small amount (usually less than half a teaspoonful) of local anaesthetic is injected into the lower back, around the nerves that go to and from the hip.

Low blood pressure is very common during surgery (at least > 30%, depending on definition), and appears to be linked to a greater chance of death within a month after surgery.

There are 2 main ways of managing low blood pressure during surgery: treatment and prevention. Treatments (fluids, drugs) have side effects in the older, frailer population with hip fracture. Prevention involves giving anaesthesia at lower doses. National guidelines recommend that lower doses are given, but this recommendation is based on historical research selectively involving younger, fitter people having hip fracture surgery. Importantly, these studies did not record blood pressure either accurately or often enough.

The Anaesthesia Sprint Audit of Practice (ASAP) 2 study suggested that a safe level of low blood pressure occurs when only 1.5 mls of spinal anaesthesia is given, and the investigator has been using this amount in Brighton since 2011. Recently, the investigator has reported a way of transferring vital signs data from anaesthetic monitors to storage computers for medicolegal purposes (e.g. in Coroner's investigations: approximately 4000 people in the UK die annually within a month of hip fracture surgery).

However, analyzing such observational data should also allow the investigator to describe accurately how blood pressure changes around the time of surgery, and in patient groups that are normally excluded from prospective research (e.g. the very old, the very frail, people with dementia). By comparing this data to published national data from the ASAP 1 study, the investigator hopes to determine whether lower doses of spinal anaesthesia are linked with a lower rate of low blood pressure during surgery, potentially improving people's survival and recovery after hip fracture.

DETAILED DESCRIPTION:
Approximately 65, 000 hip fractures occur in the UK each year, and more than 99% are repaired by surgery. Roughly half of patients receive spinal anaesthesia, where a small amount (usually ~ 2.5mls) of local anaesthetic is injected into the lower back, around the nerves that go to and from the hip.

The investigator has found that low blood pressure (hypotension) is very common during surgery (occurring in at least > 30%, depending on the definition of hypotension), and appears to be significantly linked to a greater chance of death within a month after surgery (~3% rise in mortality/5 mmHg fall in SBP).

There are 2 main ways of managing low blood pressure during surgery: treatment and prevention. Treatments (fluids, drugs) have side effects in the older, frailer population with hip fracture, including fluid overload with heart failure, and cardiac/kidney/gut ischaemia.

Prevention involves giving anaesthesia at lower doses. UK national guidelines recommend that lower doses are given (< 2mls 0.5% hyperbaric bupivacaine), but this recommendation is based on historical research selectively involving younger, fitter people having hip fracture surgery. Importantly, these studies did not record blood pressure either accurately (i.e. invasively) or often enough (i.e. > every 5 minutes).

The ASAP 2 study suggested that a safe level of low blood pressure occurs when only 1.44 mls 0.5% hyperbaric/normobaric spinal anaesthesia is administered, and the investigator has been using this amount (1.5mls) in Brighton since 2011.

Recently, it has become possible to transfer vital signs data from anaesthetic monitors to storage computers for medicolegal purposes (eg in Coroner's investigations - approximately 4000 people in the UK die annually within a month of hip fracture surgery).

However, analyzing such observational medicolegal data should also allow accurate description of how blood pressure changes around the time of surgery, and in patient groups that are normally excluded from prospective research (eg the very old, the very frail, people with dementia). By comparing this data to published national data from the ASAP 1 study, it should be possible to determine whether lower doses of spinal anaesthesia are linked with a lower rate of low blood pressure during surgery. By merging individuals' data with that held on the Brighton Hip Fracture Database, it should be possible to determine whether prevalence (and/or depth+duration of hypotension) are correlated with outcomes (survival, length of inpatient stay) after hip fracture repair.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (over 18 years) who have sustained a unilateral hip fracture and received surgery (hemiarthroplasty, dynamic hip screw, cortical screws, proximal femoral nail) under low dose spinal anaesthesia (1.3 mls 0.5% hyperbaric bupivacaine) after fascia iliaca block + sedation, administered by the Chief Investigator (CI) between 3rd March, 2017 and 1st January, 2020 at the Princess Royal Hospital, Hayward's Heath (E Sussex).
2. For whom crude vital signs data have been stored in pseudo-anonymised electronic form on secure hospital computers, for medico-legal reference

Exclusion Criteria:

1. People with hip fracture receiving conservative management during the study period;
2. People with hip fracture requiring total hip arthroplasty (for whom larger volumes of spinal anaesthesia are used);
3. People with hip fracture administered spinal anaesthesia other than 1.3 mls 0.5% hyperbaric bupivacaine;
4. People meeting inclusion criteria for whom vital signs could not be stored electronically due to equipment failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People undergoing surgical hip fracture repair (hemiarthoplasty, dynamic hip screw, cortical screws, proximal femoral nail) administered spinal anaesthesia for whom contemporaneous vital signs (including blood pressure, heart rate, oxygen saturation, breathing rate) have been stored in an anonymised, double password-protected database held on secure computers at Princess Royal Hospital, Hayward's Heath (E. Sussex).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2023-05-24 (Estimated); Study Completion 2023-05-24 (Estimated)

PRIMARY OUTCOMES:
Cohort mean (SD) mean non-invasive blood pressure (MAP) | Occurring during the 2 hour duration (approximately) of anaesthesia and surgery for each patient
  Taken at 2 minute intervals peri-operatively for each patient

SECONDARY OUTCOMES:
The cohort prevalence of hypotension | During anaesthesia and surgery
  Cohort prevalence of hypotension, variably defined as:
  1. Fall in systolic blood pressure (SBP) from baseline > 20%;
  2. Fall in systolic blood pressure (SBP) from baseline > 30%;
  3. Fall in mean arterial pressure (MAP) from baseline > 20%;
  4. Fall in mean arterial pressure (MAP) from baseline > 30%;
  5. Lowest SBP < 90 millimetres of mercury (mmHg);
  6. Lowest SBP < 100 mmHg
  7. Lowest MAP < 70 mmHg;
  8. Lowest MAP < 55 mmHg.
Mean depth x duration area under curve product for cohort hypotension after low dose spinal anaesthesia for hip fracture surgery | During anaesthesia and surgery
  Mean depth x duration area under curve product for cohort hypotension after low dose spinal anaesthesia for hip fracture surgery
Quantification of cohort systolic and mean arterial blood pressure changes before spinal administration | During anaesthesia and surgery
  Describing any effects of propofol sedation and local anaesthetic nerve block
Effective cohort duration of spinal anaesthesia | During anaesthesia and surgery
  Including number of augmentatory anaesthetic interventions required in mean (SD) time from spinal administration to surgical skin closure
Correlations between individual (a) hypotension (b) hypotension depth/duration product and outcomes (death at 30 days, length of stay in hospital) | During anaesthesia and surgery
  Correlations between individual (a) hypotension (b) hypotension depth/duration product and outcomes (death at 30 days, length of stay in hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Stu White, FRCA BSc MA, Principal Investigator — Consultant Anaesthetist
Locations (1):
- Royal Sussex County Hospital, Brighton, E Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
On application to PI
Supporting Information: Study Protocol, SAP
Time Frame: From submission for publication, indefinite
Access Criteria: Oral/written application to PI

REFERENCES:
- [Result] National Hip Fracture Database. 2019 Report. https://www.nhfd.co.uk/20/hipfractureR.nsf/docs/2019Report
- [Result] National Hip Fracture Database. Anaesthesia Sprint Audit of Practice (ASAP). 2014. https://www.nhfd.co.uk/20/hipfractureR.nsf/vwContent/asapReport/$file/onlineASAP.pdf
- [Result] White SM, Moppett IK, Griffiths R, Johansen A, Wakeman R, Boulton C, Plant F, Williams A, Pappenheim K, Majeed A, Currie CT, Grocott MP. Secondary analysis of outcomes after 11,085 hip fracture operations from the prospective UK Anaesthesia Sprint Audit of Practice (ASAP-2). Anaesthesia. 2016 May;71(5):506-14. doi: 10.1111/anae.13415. Epub 2016 Mar 4. PMID 26940645
- [Result] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Result] Ben-David B, Frankel R, Arzumonov T, Marchevsky Y, Volpin G. Minidose bupivacaine-fentanyl spinal anesthesia for surgical repair of hip fracture in the aged. Anesthesiology. 2000 Jan;92(1):6-10. doi: 10.1097/00000542-200001000-00007. PMID 10638892
- [Result] Minville V, Fourcade O, Grousset D, Chassery C, Nguyen L, Asehnoune K, Colombani A, Goulmamine L, Samii K. Spinal anesthesia using single injection small-dose bupivacaine versus continuous catheter injection techniques for surgical repair of hip fracture in elderly patients. Anesth Analg. 2006 May;102(5):1559-63. doi: 10.1213/01.ane.0000218421.18723.cf. PMID 16632842
- [Result] White SM, Pateman J. A method of recording electronic anaesthetic monitor data for research. Anaesthesia. 2017 Feb;72(2):267-269. doi: 10.1111/anae.13794. No abstract available. PMID 28093744
- [Result] White SM, Rashid N, Chakladar A. An analysis of renal dysfunction in 1511 patients with fractured neck of femur: the implications for peri-operative analgesia. Anaesthesia. 2009 Oct;64(10):1061-5. doi: 10.1111/j.1365-2044.2009.06012.x. PMID 19735395
- [Derived] White SM. A retrospective, observational, single-centre, cohort database analysis of the haemodynamic effects of low-dose spinal anaesthesia for hip fracture surgery. BJA Open. 2024 Feb 17;9:100261. doi: 10.1016/j.bjao.2024.100261. eCollection 2024 Mar. PMID 38390395